CLINICAL TRIAL: NCT03596216
Title: One-Shot Percutaneous Electrical Nerve Stimulation vs. Transcutaneous Electrical Nerve Stimulation for Performance Flexor Hallucis Longus Muscle in Professional Dancers
Brief Title: Neuromodulation in Professional Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Doctor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NM
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Rehabilitation; Sports Physical Therapy; Sport Performance; Dance
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Electrial Stimulation (PES group). (Experimental): This intervention consisted in the application of an asymmetric biphasic rectangular current. The subject lay prone with her feet outside the table. The FHL muscle was located at 50% of the distance between the fibular head and inferior border of the lateral malleolus on the posterior aspect of the fibular by ultrasound machine (cross-section) (Logiq, GE Healthcare, USA) and then, a needle (0.30mm x 0.40mm) was inserted, perpendicular to the surface of the skin, until the muscle belly. Prior to inserting a neddle, the underlying skin was cleaned with isopropyl alcohol. The intensity of the current was necessary to cause an exacerbated muscle contraction, during 1.5 min acording to the Valera and Minaya protocol´s.
  This intervention was performed once in each participant, on one leg only (stance limb), It's only once, it was not a treatment
  Interventions: Other: PENS
- Transcutaneous Electrial Stimulation (TENS group) (Experimental): This intervention consisted in the application of an asymmetric biphasic rectangular current. The subject lay prone with her feet outside the table. The FHL muscle was located at 50% of the distance between the fibular head and inferior border of the lateral malleolus on the posterior aspect of the fibular by ultrasound machine (cross-section) (Logiq, GE Healthcare, USA),and then, one self-adhesive electrode was placed on the back of the leg and the other on the sole of the foot. The intensity of the current was necessary to cause an exacerbated muscle contraction, during 1.5 min.
  This intervention was performed once in each participant, on one leg only (stance limb), It's only once, it was not a treatment
  Interventions: Other: TENS

INTERVENTIONS:
Other: PENS — This intervention consisted in the application of an asymmetric biphasic rectangular current of 150 microseconds and 10 Hz using a specifically developed medically certified device (Physio Invasive, Enraf Nonius, Prim, SPAIN). This is an invasive intervention by ultrasound and needles.
  Arms: Percutaneous Electrial Stimulation (PES group).
Other: TENS — This intervention consisted in the application of an asymmetric biphasic rectangular current of 150 microseconds and 10 Hz using a specifically developed medically certified device (Physio Invasive, Enraf Nonius, Prim, SPAIN). This is a non-invasive intervention by self-adhesive electrodes.
  Arms: Transcutaneous Electrial Stimulation (TENS group)

SUMMARY:
Tendinopathy of the flexor hallucis longus (FHL), colloquially referred to as "dancer's tendinitis," is a common condition in dancers and attributed to high demand on this muscle in positions of extreme ankle plantarflexion and metatarsophalangeal (MTP) flexion and extension. Tradicional conservative treatment includes rest from pain-inducing activities including pointe work and jumping, physical therapy a focusing on movilization of the joints of the first ray and subtalar joint, and antiinflamatory medications. Unfortunately, dancer frecuently do not follow recommendations to rest due to the competitive nature of the field. Those who do not respond to conservative treatment undergo more serious interventions including steroid injections or surgery, each with additional risks and recovery time. To develop experimental protocols aimed at prevention and nonsurgical interventions are needed. Therefore, the aim of this study was To investigate the effects of one shot of low-frequency percutaneous electrical nerve stimulation (PENS) vs. one shot of transcutaneous electrical nerve stimulation (TENS) in performance of the Flexor Hallucis Longus muscle in young dancers.

ELIGIBILITY:
Inclusion Criteria:

* Female dancers
* Training at least twenty-five hours per week
* Pointe training at least five hours per week.

Exclusion Criteria:

* They had sustained an injury to their stance limb in the past year preventing dancing for at least 1 day
* Personal Psychological Apprehension Scale (PPAS) score >37.5
* Commonly accepted contraindications to invasive phsyiotherapist technique
* Any contraindications to needling per se.
* Commonly accepted contraindications to electrotherapy
* Epilepsy.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Change in balance | 1 day
  Assessed by a single leg balance test
Change in muscular endurence, | 1 day
  Assessed by endurance test (heel raise repetitions).
Change in range of motion of first MTF joint | 1 day
  Assessed using goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca De la Cruz Torres, Dr, Study Chair — University of Seville
Locations (1):
- Blanca de La Cruz Torres, Seville, Spain

REFERENCES:
- [Background] de-la-Cruz-Torres B, Barrera-Garcia-Martin I, Romero-Morales C. Comparative Effects of One-Shot Electrical Stimulation on Performance of the Flexor Hallucis Longus Muscle in Professional Dancers: Percutaneous Versus Transcutaneous? Neuromodulation. 2020 Aug;23(6):865-870. doi: 10.1111/ner.13040. Epub 2019 Aug 25. PMID 31448488